CLINICAL TRIAL: NCT04791111
Title: AQUA: A NEW QUESTIONNAIRE ASSESSING ANTICHOLINERGIC SIDE EFFECTS IN NEUROGENIC POPULATION (AQUA: Anticholinergic Side Effects QUestionnAire)
Brief Title: AQUA: Anticholinergic Side Effects QUestionnAire
Acronym: AQUA
Status: Completed | Type: Observational
Sponsor: Pierre and Marie Curie University (Other)
Responsible Party: Principal Investigator, Gérard Amarenco, Clinical professor, Head of neuro urology department, APHP, tenon Hospital, Paris, France, Pierre and Marie Curie University
Other Study IDs: GREEN GRC-01
Record Dates: First submitted 2021-03-05; First posted 2021-03-10 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Overactive Bladder
Keywords: tool; side effects; questionnaire; neurogenic bladder
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Bladder, Neurogenic | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — validated questionnaire to assess side effects secondary to antimuscarinics treatment in neurogenic bladder

SUMMARY:
Overactive bladder syndrome (OAB) is very frequent and increase with age. Antimuscarinics allows improvement for OAB symptoms, quality of life and urodynamic parameters. However, antimuscarinics adherence is poor and anticholinergic drugs are often withdrawn few months after their introduction. This low adherence to antimuscarinics can be explained by side effects as dry mouth, blurred vision, constipation or cognitive impairment which are due to systemic anticholinergic effects since specificity and receptor affinity of bladder antimuscarinics are poor with a large distribution of acetylcholine receptors in all the body. Unfortunately, there is no questionnaires which evaluate side effects or constraints. The objective of the study is to develop and validate a new questionnaire to assess side effects of antimuscarinic treatment in a patient with OAB.

The study was conducted in a Neuro-urology Department of a University Hospital. To allow a full psychometric validation of the questionnaire, the study protocol included 3 steps: qualitative interviews, feasibility study and validation study. The inclusion criteria were to be aged > 18 years and to have OAB symptoms according to the ICS definition and secondary to a neurogenic dysfunction.

First step of the study consisted in a review literature on Pubmed to explore the different side effects secondary to antimuscarinic treatment and do determine which tools were available. In addition, we conducted semi-structured interviews on 30 patients suffering from OAB.

For this feasibility study, 30 patients were included. They had to rate each item to evaluate comprehension, acceptation and pertinence with a three-points Likert scale from response "0: not at all or quite" to "2: perfectly".

Validation study: 100 patients Content validity was assessed by the panel of experts. Internal consistency reliability was calculated using the α coefficient of Cronbach. Each response has been transformed in a numeric value to perform this test. Alpha coefficient of Cronbach was considered as very good if > 0.7.

Test-retest reliability was tested using the intraclass correlation coefficient (ICC) which was significant over 0.7.

Objective was to validate this questionnaire with good or very good psychometric properties. Primary outcome was Alpha coefficient of Cronbach and ICC ≥ 0,7.

DETAILED DESCRIPTION:
Lower Urinary tract symptoms (LUTS) are widespread in the general population and their prevalence is expected to increase in the coming years as the elderly population increases. Indeed, overactive bladder syndrome (OAB) is very frequent and increase with age. OAB has numerous and various etiologies and can be caused by urologic, metabolic, neurogenic or autonomic dysfunction. Treatments for OAB depends on etiology but first line treatment often corresponds to lifestyle modification and antimuscarinics. Antimuscarinics allows improvement for OAB symptoms, quality of life and urodynamic parameters. However, antimuscarinics adherence is poor and anticholinergic drugs are often withdrawn few months after their introduction. This low adherence to antimuscarinics can be explained by side effects as dry mouth, blurred vision, constipation or cognitive impairment which are due to systemic anticholinergic effects since specificity and receptor affinity of bladder antimuscarinics are poor with a large distribution of acetylcholine receptors in all the body. Unfortunately, there is no or a few questionnaires which evaluate side effects or constraints, except for one published in 2019, but not specific for anticholinergics. This part of evaluation is poorly reported in medical literature, whereas it seems to be clear that side effects should be systematically evaluate and are in part responsible of treatment discontinuation. The objective of the study is to develop and validate a new questionnaire to assess side effects of antimuscarinic treatment in a patient with OAB.

The study was conducted in a Neuro-urology Department of a University Hospital. To allow a full psychometric validation of the questionnaire, the study protocol included 3 steps: qualitative interviews, feasibility study and validation study. The inclusion criteria were to be aged > 18 years and to have OAB symptoms according to the ICS definition and secondary to a neurogenic dysfunction.

First step of the study consisted in a review literature on Pubmed to explore the different side effects secondary to antimuscarinic treatment and do determine which tools were available. In addition, we conducted semi-structured interviews on 30 patients suffering from OAB.

Feasibility Study For this feasibility study, 30 patients were included. They had to rate each item to evaluate comprehension, acceptation and pertinence with a three-points Likert scale from response "0: not at all or quite" to "2: perfectly".

Validation study: 100 patients Content validity was assessed by the panel of experts. Internal consistency reliability was calculated using the α coefficient of Cronbach. Each response has been transformed in a numeric value to perform this test. Alpha coefficient of Cronbach was considered as very good if > 0.7.

Test-retest reliability was tested using the intraclass correlation coefficient (ICC) which was significant over 0.7. The first questionnaire was filled at the end of the first consultation and patients had to answer a second questionnaire (filled at home) 7 days after the first consultation.

Objective was to validate this questionnaire with good or very good psychometric properties. Primary outcome was Alpha coefficient of Cronbach and ICC ≥ 0,7.

ELIGIBILITY:
Inclusion Criteria:

* OAB symptoms according to ICS definition
* neurogenic bladder
* antimuscarinic treatment

Exclusion Criteria:

* Treatment change between first evaluation and second evaluation (Test retest validity)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient suffering from OAB symptoms secondary to neurogenic condition and treated by antimuscarinic treatment.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
reproductibilty of Anticholinergic side effects QuestionnAire (AQUA) | 1 day
  Patients were asked to answer a second time the questionnaire with a second evaluation at 14 days after the first one. The "intra-class correlation coefficient" (ICC) was used to detemrine if this evaluaiton could lead to similar result for each quesiton. An ICC>0.70 was necessary to define reproductibility.
Acceptatbility of AQUA | 1 day
  Each patient was asked to rate acceptatibilty of the questionnaire with a four-point liket scale (A: perfect, B : good, C: Average, D: bad) regarding acceptance of the questions
Comprehension of AQUA | 1 day
  Each patient was asked to rate comprehension of the questionnaire with a four-point liket scale (A: perfect, B : good, C: Average, D: bad) regarding comprehension of the questions

CONTACTS AND LOCATIONS:
Overall Officials: Gérard AMARENCO, MD, PhD, Principal Investigator — Sorbonne University, GRC 001, GREEN, APHP, Hopital Tenon, France
Locations (1):
- department of Neuro-Urology, Hôpital Tenon, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided